CLINICAL TRIAL: NCT07339345
Title: Prospective Single-Arm Clinical Trial of Golidocitinib Monotherapy for Hemophagocytic Lymphohistiocytosis.
Brief Title: Prospective Single-Arm Clinical Trial of GO Regimen for HLH.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Doctor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Golidocitinib(GO),HLH
Record Dates: First submitted 2026-01-01; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Lymphohistiocytosis, Hemophagocytic
Keywords: Hemophagocytic Lymphohistocytosis; Golidocitinib
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLH patients (Experimental): Initial diagnosis or presence of refractory/relapsed HLH disease or confirmed diagnosis of HLH.
  Interventions: Drug: Golidocitinib

INTERVENTIONS:
Drug: Golidocitinib — Administer the GO regimen to HLH patients who meet the inclusion criteria, specifically Golicitinib 150 mg once daily.

SUMMARY:
This study aims to investigate the efficacy and safety of Golidocitinib(GO) monotherapy in the treatment of hemophagocytic lymphohistiocytosis.

ELIGIBILITY:
Inclusion Criteria:

1. Researchers evaluate patients with newly diagnosed or refractory/relapsed HLH disease.
2. Definite diagnosis of HLH: molecular diagnosis consistent with pHLH, or at least 5 of the 8 criteria in the HLH-2004 diagnostic criteria.
3. Patients who are currently unsuitable or unable to undergo allo-HSCT.
4. Researchers estimate that the expected survival period exceeds one month.
5. Patients must be at least 14 years of age and no older than 70 years of age, with no gender restrictions.
6. Before the study began, TB was ≤10 times the upper limit of normal; Cr was ≤1.5 times the normal value.
7. Serum HIV antigen or antibody negative。
8. HCV antibody negative, or HCV antibody positive but HCV RNA negative.
9. .HBsAg and HBcAb are both negative. If either of the above is positive, peripheral blood hepatitis B virus DNA titer testing is required, with a titer of less than 1×10³ copies/ml.
10. Echocardiography showed LVEF ≥ 50%.
11. Women of childbearing age must be confirmed as not pregnant by a pregnancy test and must be willing to use effective contraception during the study period and for at least 12 months after the last dose; all male participants must use contraception during the study period and for at least 3 months after the last dose.

Exclusion Criteria:

1. Heart function above grade II(including II) (NYHA).
2. Pregnancy or lactating Women and reproductive-age patients who refused to use appropriate contraceptive measures during this trial.
3. Individuals who are allergic to GO or have a severe allergic constitution.
4. Active bleeding of the internal organs.
5. uncontrollable infection.
6. Severe mental illness.
7. History of non-melanoma skin cancer.
8. Unable to comply during the trial and/or follow-up phase. Participate in other clinical research at the same time.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2027-06-27 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment response | Weeks 2, 4, 6, and 8 after the start of treatment
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, triglyceride, blood cell count, hemophagocytosis, and level of consciousness (if CNS HLH is present).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; without blood transfusion: Neutrophils <500/ml must increase by 100% and be >500/ml; neutrophils 500-2000/ml must increase by 100% and return to normal.; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.
  No response is defined as not meeting the criteria for partial response.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 days after the last dose is administered.
  An adverse event is defined as an adverse medical condition (including worsening of a pre-existing condition) that occurs in a subject or clinical trial subject after receiving medication, regardless of whether it is causally related to the investigational drug.
  Serious adverse events are defined as AEs that meet one or more of the following criteria during any study period: death; immediate threat to life; and hospitalization or prolongation of hospitalization.

OTHER OUTCOMES:
Survival | 1 year
  Patient's HLH-related symptoms and auxiliary examination results

CONTACTS AND LOCATIONS:
Overall Officials: zhao Wang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China